CLINICAL TRIAL: NCT06263829
Title: Effectiveness of a Novel Smart Tag Technology in a Pharmacy-Led Setting to Improve Adherence, Patient-Centered Care and Outcomes in HCV
Brief Title: HCV Tappt Adherence Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Synchronyx (Unknown); American Society of Health-System Pharmacists (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-1580
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tappt App (Experimental): Participants will download and utilize the Tappt app to record adherence to oral medication. For the purposes of this study, adherence for participants in the intervention arm will be measured using a modified medication possession ratio (MPR) measure called medication tag scan ratio (MTSR). MTSR is defined as a percentage of the number of times participants scanned their passive tags versus the total of expected tag scans based on that participant's medication regimen and treatment period.
  Interventions: Other: Use of Tappt App
- Historical Control (No Intervention): Upon study completion, a retrospective matched control will be established for the intervention group. Historic data for the matched control's adherence, treatment completion, SVR assessment, and SVR rates will be compared to the intervention arm.

INTERVENTIONS:
Other: Use of Tappt App — Use of Tappt, a novel digital medication companion solution
  Arms: Tappt App

SUMMARY:
The goal of this non-inferiority clinical trial is to evaluate the efficacy of Tappt, a novel digital medication companion solution, among individuals with hepatitis C virus (HCV) who are starting a daily oral medication regimen following standard of care in a clinical pharmacy setting.

* The primary aim is to assess the non-inferiority of Tappt with medication adherence, treatment completion, sustained virologic response (SVR) assessment, and SVR achievement rates.
* The secondary aim is to assess the efficacy of Tappt at enabling pharmacists to personalize treatment and management decision based on participants' reported barriers to adherence, care, and SVR achievement.

Participants will download and utilize the Tappt app to record adherence to oral medication. For the purposes of this study, adherence for participants in the intervention arm will be measured using a modified medication possession ratio (MPR) measure called medication tag scan ratio (MTSR). MTSR is defined as a percentage of the number of times participants scanned their passive tags versus the total of expected tag scans based on that participant's medication regimen and treatment period.

Upon study completion, a retrospective matched control will be established for the intervention group. Historic data for the matched control's adherence, treatment completion, SVR assessment, and SVR rates will be compared to the intervention arm.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Hepatitis C virus (HCV) infection (denoted by positive HCV antibody and detectable HCV RNA)
3. Initiating oral HCV therapy with glecaprevir/pibrentasvir or sofosbuvir/velpatasvir
4. HCV treatment provided and managed by the clinical pharmacist at UI Health
5. Access to a mobile smartphone (iPhone 7 or later; Android release date 2012 or later) with reliable data and/or Wi-Fi access
6. Ability to verbalize understanding of the study protocol in English
7. Able and willing to provide informed consent in English

Exclusion Criteria:

1. Inability to speak and read English
2. Inability or unwillingness to adhere to the study protocol
3. Pregnant individuals
4. Decompensated cirrhosis (Child Turcotte Pugh Class B and C); hepatocellular carcinoma; prior liver or kidney transplant

No patient will be excluded because of gender, race or ethnic origin.

The following populations will be excluded from the study:

* Adults 18 years of age and older who are unable or unwilling to consent
* Individuals less than 18 years old
* Pregnant individuals
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | 8-12 weeks
  Modified medication possession ratio (MPR) measure called medication tag scan ratio (MTSR)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Martin, Principal Investigator — UIH
Locations (1):
- UIH, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.